CLINICAL TRIAL: NCT02177630
Title: Myocarditis and the Role of Advanced Magnetic Resonance Imaging
Brief Title: Magnetic Resonance Imaging in Myocarditis
Acronym: MyoRacer
Status: Completed | Type: Observational
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Other Study IDs: 123456123456
Record Dates: First submitted 2014-06-22; First posted 2014-06-27 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Myocarditis
Keywords: myocarditis, myocardial inflammation, imaging, magnetic resonance
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Magnetic resonance imaging and endomyocardial biopsy: Magnetic resonance imaging and endomyocardial biopsy
  Interventions: Other: Endomyocardial Biopsy

INTERVENTIONS:
Other: Endomyocardial Biopsy

SUMMARY:
The purpose of this study is the assess the diagnostic performance of magnetic resonance imaging in patients with suspected myocarditis by applying different imaging sequences at different MR scanners

DETAILED DESCRIPTION:
In patients with clinical suspicion of myocarditis biventricular endomyocardial biopsy is performed for definite diagnosis. In addition, patients undergo magnetic resonance imaging at 1.5 Tesla and 3.0 Tesla within 24 hours. The imaging protocol of both scan include assessment of myocardial edema respectively edema ratio; myocardial hyperemia respectively global relative enhancement (gRE); myocardial fibrosis/necrosis respectively myocardial LE and T1 and T2 mapping sentences. Diagnostic performance of different imaging protocols as compared to the findings of endomyocardial biopsies is calculated.

The protocol also includes a follow-up MR can at 3 months.

ELIGIBILITY:
Inclusion Criteria:

Symptoms such as:

* Dyspnea or Orthopnea or
* Palpitations or
* Exercise intolerance or
* Angina

Evidence of myocardial involvement:

* ventricular dysfunction on echocardiography or
* new or persistent ECG changes
* elevated Troponin T History of viral infection

Exclusion Criteria:

* Contraindication for magnetic resonance imaging
* Impaired renal function: glomerular filtration rate ≤ 30 ml/min/m2
* Patients presenting with pregnancy
* Patients without informed consent
* Participation in another trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical suspicion of myocarditis
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Accuracy, sensitivity and specificity of magnetic resonance imaging sequences | baseline
  The diagnostic accuracy of individual and a combination of MR imaging sequences (late enhancement images, assessment of global edema, relative enhancement and T1 and T2 mapping sequences) will be determined by comparison to endomyocardial biopsies, which serve as diagnostic gold-standard

SECONDARY OUTCOMES:
Diagnostic performance of biventricular endomyocardial biopsies | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lurz, MD, PhD, Principal Investigator — Heart Center of the University of Leipzig
Locations (1):
- Heart Center of the University Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Baessler B, Luecke C, Lurz J, Klingel K, Das A, von Roeder M, de Waha-Thiele S, Besler C, Rommel KP, Maintz D, Gutberlet M, Thiele H, Lurz P. Cardiac MRI and Texture Analysis of Myocardial T1 and T2 Maps in Myocarditis with Acute versus Chronic Symptoms of Heart Failure. Radiology. 2019 Sep;292(3):608-617. doi: 10.1148/radiol.2019190101. Epub 2019 Jul 30. PMID 31361205
- [Derived] Lurz P, Luecke C, Eitel I, Fohrenbach F, Frank C, Grothoff M, de Waha S, Rommel KP, Lurz JA, Klingel K, Kandolf R, Schuler G, Thiele H, Gutberlet M. Comprehensive Cardiac Magnetic Resonance Imaging in Patients With Suspected Myocarditis: The MyoRacer-Trial. J Am Coll Cardiol. 2016 Apr 19;67(15):1800-1811. doi: 10.1016/j.jacc.2016.02.013. PMID 27081020